CLINICAL TRIAL: NCT02003287
Title: Determining the Efficacy of Using FEES Compared to VFSS to Diagnose Laryngeal Penetration and Aspiration in Infants in the Neonatal Intensive Care Unit (NICU)
Brief Title: Comparing FEES to VFSS in Diagnosing Laryngeal Penetration and Aspiration in Infants in the NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 012-282
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Deglutition Disorders
Keywords: Deglutition Disorders; Intensive Care Units, Neonatal
MeSH Terms: conditions — Deglutition Disorders | interventions — Fees and Charges

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FEES (Experimental): Swallowing evaluation with the Fiberoptic Endoscopic Evaluation of Swallowing
  Interventions: Other: FEES
- VFSS (Active Comparator): Swallowing evaluation with the Videofluoroscopic Swallowing Study
  Interventions: Other: VFSS

INTERVENTIONS:
Other: VFSS — Videofluoroscopic Swallow Study
  Arms: VFSS
Other: FEES — Fiberoptic Endoscopic Swallow Study
  Arms: FEES

SUMMARY:
The main purpose of the study is to determine whether the Fiberoptic Endoscopic Evaluation of Swallowing (FEES) is effective in detecting laryngeal penetration and tracheal aspiration when compared with the Videofluoroscopic Swallowing Study (VFSS) in bottle-feeding infants in the NICU. A secondary objective is to determine whether FEES can be used to detect laryngeal penetration and tracheal aspiration in breastfeeding NICU infants.

ELIGIBILITY:
Inclusion Criteria:

* 37 weeks or more postmenstrual age
* Diagnosis or suspicion of laryngeal penetration and/or tracheal aspiration by neonatal therapist and/or physician
* Inpatient at Baylor University Medical Center NICU

Exclusion Criteria:

* Not medically stable enough to undergo both FEES and VFSS as determined by neonatal therapist and/or physician
* Bilateral complete cleft lip and palate

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
High sensitivity and specificity values for FEES | one year

SECONDARY OUTCOMES:
Evidence of laryngeal penetration or tracheal aspiration during breastfeeding | at time of assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa S. Suterwala, M.D., Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] da Silva AP, Lubianca Neto JF, Santoro PP. Comparison between videofluoroscopy and endoscopic evaluation of swallowing for the diagnosis of dysphagia in children. Otolaryngol Head Neck Surg. 2010 Aug;143(2):204-9. doi: 10.1016/j.otohns.2010.03.027. PMID 20647120
- [Background] Leder SB, Karas DE. Fiberoptic endoscopic evaluation of swallowing in the pediatric population. Laryngoscope. 2000 Jul;110(7):1132-6. doi: 10.1097/00005537-200007000-00012. PMID 10892683
- [Derived] Suterwala MS, Reynolds J, Carroll S, Sturdivant C, Armstrong ES. Using fiberoptic endoscopic evaluation of swallowing to detect laryngeal penetration and aspiration in infants in the neonatal intensive care unit. J Perinatol. 2017 Apr;37(4):404-408. doi: 10.1038/jp.2016.239. Epub 2017 Jan 5. PMID 28055025